CLINICAL TRIAL: NCT02373111
Title: Effects of Isoflavone Combined With Astaxanthin on Skin Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Ho Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-1412-144-637
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Ageing; Photo-aging
Keywords: Anti-aging; Isoflavones; Astaxanthine; Skin aging
MeSH Terms: interventions — Isoflavones; astaxanthine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isoflavone and Astaxanthin (Active Comparator): Each subject takes one active tablet per day for 24 weeks. Each tablet contains isoflavone 27mg and astaxanthin 4mg.
  Interventions: Dietary Supplement: Isoflavone; Dietary Supplement: Astaxanthin
- Placebo (Placebo Comparator): Each subject takes one placebo tablet per day for 24 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Isoflavone
  Arms: Isoflavone and Astaxanthin
Dietary Supplement: Astaxanthin
  Arms: Isoflavone and Astaxanthin
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Photoaging is caused by the superposition of chronic ultraviolet (UV)-induced damage on the intrinsic aging process, and accounts for the majority of age-associated changes in skin appearance. Reactive oxygen species (ROS) play a key role in UV-induced skin damage and diminish skin matrix protein levels, leading skin aging. Strategies utilizing endogenous skin antioxidants as well as plant-derived or synthetic compounds have been examined.

Astaxanthin mainly from marine algae and crustaceans is a kind of carotenoids which were well-known photo-protective agents with strong antioxidant activity. Several studies have revealed that supplementation of astaxanthin effectively protect skin against UV damage through free radicals.

In addition, matrix metalloproteinase-1 induced by UV irradiation is an important step toward skin aging. Recently, many studies pointed out that phytoestrogens exhibit agonistic and antagonistic estrogen activities, suppressing activity of MMP-1 in skin. Isoflavone is a kind of phytoestrogen from soybean and mainly act on skin and bones, inhibiting MMP-1 effectively.

The present study is designed to take isoflavone combined with astaxanthin to maximize their anti-aging ability and objectively measure the effects of the mixture on facial wrinkles, hydration, and elasticity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females aged ≥ 45 years
* Facial wrinkle grade 2 to 4

Exclusion Criteria:

* received medical or cosmetic treatment that interferes with the general aging process at least 3 months before the study
* received any hormone replacement therapy at least 3 months before the study
* reported taking functional foods more than 1 month during last 3 months before the study
* history of acute or chronic disease such as severe liver or kidney disease
* history of allergies against any component of trial foods
* any visible skin disease that might be confused with a skin reaction to the test procedure

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in skin wrinkles | Twenty-four weeks
  Facial wrinkles in the crow's feet area measured by Skin Visiometer

SECONDARY OUTCOMES:
Change from baseline in skin elasticity | Twenty-four weeks
  Facial elasticity measured by Cutometer
Change from baseline in epidermal hydration | Twenty-four weeks
  Skin hydration measured by Corneometer
Change from baseline in skin barrier integrity | Tewnty-four weeks
  TEWL measured by Tewameter

CONTACTS AND LOCATIONS:
Overall Officials: Jin Ho Chung, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea